CLINICAL TRIAL: NCT00645112
Title: A Comparison of Safety and Efficacy of Cefdinir Oral Suspension Versus Azithromycin in Pediatric Subjects With Acute Otitis Media
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, Abbott
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M03-630
Record Dates: First submitted 2008-03-22; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Cefdinir; Azithromycin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cefdinir (Omnicef)
- 2 (Active Comparator)
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: cefdinir (Omnicef) — oral suspension, 7 mg/kg every 12 hours for 5 days
  Other Names: ABT-198; Omnicef; cefdinir
  Arms: 1
Drug: azithromycin — oral suspension 10 mg/kg QD on Day 1 then 5 mg/kg QD on Days 2-5 for a total of 5 days.
  Arms: 2

SUMMARY:
To compare the safety and efficacy of cefdinir oral suspension, 7 mg/kg every 12 hours for 5 days, to azithromycin oral suspension 10 mg/kg/day (Day 1) then 5 mg/kg/day (Days 2-5) for a total of 5 days, in children between 6 months and 6 years of age, with AOM.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, documented by medical history and physical examination, is AOM I 1 week.
* Clinical symptoms include >=1 of the following: Otalgia (earache or pain), this may be expressed as ear pulling or nabbing; Ear fullness; Decreased hearing, this may be based on reports from parents or legally authorized representatives; Discharge from the external auditory canal (following acute perforation of the tympanic membrane).
* At least two (2) of the following signs are present in at least one ear: Full or bulging or perforated tympanic membrane, which may be erythematous (note - since hyperemia may be present in a febrile or crying child, a red tympanic membrane alone is insufficient for the diagnosis of AOM); Loss of tympanic membrane landmarks (opacity of the tympanic membrane); Abnormal tympanic membrane mobility on biphasic pneumatic otoscopy, due to the presence of pus or fluid behind the tympanic membrane and edema of the tympanic membrane. Have evidence of middle ear fluid demonstrated by acoustic reflect tympanometry (ear check) showing values of 3, 4 or 5.
* Generally in good health based on medical history, vital signs, physical exam, and historical laboratory results.
* Subject must be a suitable candidate for oral antibiotic therapy.

Exclusion Criteria:

* Previous enrollment in this study.
* Enrollment in any other investigational study using unapproved products or unapproved doses; in the previous four weeks prior to study start.
* Hypersensitivity reactions to cefdinir, other cephalosporins, azithromycin, other macrolide and azalide antibiotics, and/or sensitivity to multiple allergens.
* Presence of tympanostorny tubes or otitis externa at Evaluation 1.
* Systemic treatment with any anti-infective agent within 14 days prior to Evaluation 1 or during the study.
* Treatment with a long-acting injectable antimicrobial agent (e.g., penicillin G benzathine) within 4 weeks prior to study drug administration.
* Concomitant infection that requires additional antimicrobial therapy.
* Evidence of chronic, suppurative otitis media.
* Evidence of perforation of the tympanic membrane > 24 hours.
* Evidence of a physiologic, anatomic, or immunologic defect, which would interfere with resolution of this episode of acute otitis media.
* Immunocompromised subject (e.g., neutropenic subjects).
* Presence of a disease, complicating factor (e.g., mastoiditis), or structural abnormality that would preclude evaluation of the subject's therapeutic response.
* Any expectation that treatment with probenecid will be expected during the study drug administration period.
* Known significant renal or hepatic impairment.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 357 (Actual)
Dates: Start 2003-11; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate at Evaluation 2 | 9 days

SECONDARY OUTCOMES:
Sustained clinical cure rate at Evaluation 4 | 25 days

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Columbiana, Alabama
  - Montgomery, Alabama
  - Ozark, Alabama
  - Fresno, California
  - Marietta, Georgia
  - Stone Mountain, Georgia
  - Dubuque, Iowa
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Cadillac, Michigan
  - Kalamazoo, Michigan
  - Portage, Michigan
  - Richland, Michigan
  - Omaha, Nebraska
  - Columbus, Ohio
  - Huber Heights, Ohio
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Sellersville, Pennsylvania
  - Charleston, South Carolina
  - Kingsport, Tennessee
  - Lake Jackson, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Vienna, Virginia
  - Monroe, Wisconsin